CLINICAL TRIAL: NCT03750435
Title: ZERO Radiation Exposure for Catheter Ablation of Atrial Fibrillation or Left Atrial Tachycardia
Brief Title: Non-fluoroscopy Ablation of AF/AT
Acronym: ZERO-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Baylis Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMRBH01
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: AF - Atrial Fibrillation; Atrial Tachycardia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: prospective single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation for AF or left-sided AT (Experimental): The patient will be admitted in hospital as for a standard ablation procedure and discharged the next day. The procedure will be carried out without using fluoroscopy and relying on the visualization of the electroanatomical mapping system.
  Interventions: Procedure: AF ablation or left-sided AT ablation

INTERVENTIONS:
Procedure: AF ablation or left-sided AT ablation — According to the type of AF/AT, single or double transseptal and subsequent catheter ablation in the left atrium using radiofrequency will be performed.

SUMMARY:
Atrial fibrillation is the most common arrhythmia but can be treated by a catheter procedure where specialized wires (so-called catheters) are inserted in the left upper heart chamber. This requires crossing the wall between the right and left atrium with a long needle (a so-called transseptal puncture or TSP). This is typically done using x-ray guidance or echo to check if the needle is in the right position. The investigators developed a method to do the TSP without x-rays using a specialized needle that can be also shown as a little icon on the 3D electroanatomical mapping system (CARTO).3D mapping systems are routinely used to track the location of the catheters in cath labs worldwide, but the position of the needle was not tracked yet. The investigators seek to demonstrate that these procedures can be carried out safely, successfully and in a reproducible fashion without any radiation by taking advantage of "faking" the isolated tip of the needle as a catheter on the 3D mapping system. The results will be compared with historic procedures done by the same operator in the years 2012-2017.

DETAILED DESCRIPTION:
The hypothesis is that patients who undergo one or more TSP(s) for atrial fibrillation or left atrial tachycardia can be studied without the use of fluoroscopy which should result in a low or ZERO overall radiation exposure for the entire ablation procedure. The investigators will assess the feasibility, safety and efficacy of this new approach.

The patient will be admitted in hospital as for a standard procedure and discharged the next day. Before admission, the patient undergoes a CMR/CT scan (routine in our centre). To avoid total radiation CMR would be preferred, if possible.

The technique of the TSP and the use of the RF needle is commonly used worldwide. The ability to visualize the needle tip on the 3D electroanatomical mapping system facilitates the procedure. The additional visualization by TOE helps to assure that the fossa ovalis has been correctly identified.

After the TSP, the ablation procedure itself will be carried out as conventionally performed using the catheter visualization on the 3D mapping system.

An ECG and an echocardiogram are performed before discharge (as standard care).

At 3 months the patient comes for the first visit and has an ECG, a Holter and symptom questionnaire.

At 6 months, the patient has second visit which includes an ECG, a symptom questionnaire, a Holter and an echocardiogram.

If recurrences of any arrhythmia occur, the patient can be scheduled for a second ablation procedure without any restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Any type of atrial fibrillation or left atrial tachycardia

  * Able to give written informed consent
  * Age >18 years old and ≤ 80 years
  * Fulfill established clinical criteria for catheter ablation of atrial fibrillation (1)
  * No evidence of significant structural heart disease or congenital heart disease

Exclusion Criteria:

Intolerance or unwillingness to oral anticoagulation with Warfarin

* Bleeding disorder
* Contraindication to CT scan
* Presence of intracardiac thrombus
* Vascular disorder preventing access to femoral veins
* Cardiac congenital abnormality
* Severe, life threatening non-cardiac disease
* Active malignant disease and recent (<5 years) malignant disease
* Presence of ASD or PFO closure device
* Unable or unwilling to comply with F/U requirements
* Renal impairment
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-08 (Estimated)

PRIMARY OUTCOMES:
Safety of the zero AF procedure | 6 months
  Absence of acute adverse events due to the use of non-fluoroscopic AF ablation
  • Evidence of chronic adverse events due to the use of non-fluoroscopic catheter ablation during the 6 months F/U period
Feasibility and efficacy | 6 months
  Assessment on efficacy of non-fluoroscopic AF acutely and if recurrences in 6 months follow up

SECONDARY OUTCOMES:
Recurrences | 6 months
  * Time to first recurrence of AF/flutter/tachycardia (>30 sec)
  * Freedom of AF on previously failed antiarrhythmic medication; time-dependant variable
  * AF/flutter/tachycardia (> 30 sec) burden at 6 months F/U; this will be modelled as a continuous variable (number of episodes recorded)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Ernst, MD, Principal Investigator — Royal Brompton and Harefield NHS; Sabine Ernst, MD, Study Director — Royal Brompton and Harefield NHS
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Any data of this trial will be shared only in an anonymised fashion and as part of scientific publications